CLINICAL TRIAL: NCT03028025
Title: Radial Hemostasis is Facilitated With a Potassium Ferrate Hemostatic Patch (Statseal): the Randomized Controlled Statseal With TR Band Assessment Trial (STAT)
Brief Title: Comparing TR Band to Statseal in Conjunction With TR Band
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Long Beach Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arnold Seto, Chief of Cardiology, VA Long Beach Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MIRB 1427
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Arterial Occlusion; Angina Pectoris; Cardiovascular Diseases; Atherosclerosis; Hematoma; Anticoagulant-Induced Bleeding; Coronary Artery Disease
Keywords: radial artery occlusion; time to hemostasis; radial artery; transradial catheterization; TR band; Statseal; hemostasis band; potassium ferrate; percutaneous coronary intervention
MeSH Terms: conditions — Arterial Occlusive Diseases; Angina Pectoris; Cardiovascular Diseases; Atherosclerosis; Hematoma; Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TR Band Only (Active Comparator): TR Band: Patients randomly assigned to the control group will have a TR band applied over the arteriotomy site and inflated with 15-18ml of air. After aspirating and clearing the contents of the sheath, the radial sheath will be removed. The TR band will be deflated until bleeding occurs, and 2 ml of air will be reintroduced to provide hemostasis. Patent hemostasis will be documented with plethysmography and oximetry as described below within 5 minutes after band application and removal, and within 30 min of discharge or after 24 hours. The TR band will be left inflated and in place for 2 hours following the procedure for all patients (regardless of diagnostic or PCI procedure), after which deflation attempts will commence.
  Interventions: Device: TR Band
- Statseal with TR Band (Experimental): StatSeal: Patients randomly assigned to the experimental group will have a Statseal Advance (SSA) disc applied after withdrawing the radial sheath 2-4 cm. A Tegaderm dressing will be applied to secure the disc position. The TR band will be applied over the SSA disc with the center of the balloon (the green dot) over the center of the SSA disc. The TR band will be inflated with 8cc of air (which is typically occlusive pressure), and the sheath removed. No deflation will occur immediately. After 20 minutes of pressure, 3 cc of air will be removed from the TR band. After an additional 20 minutes (40 minutes after procedure), the TR band will be completely deflated, and the TR band left in place. After an additional 20 minutes (60 minutes after procedure) the TR band will be removed.
  Interventions: Device: StatSeal

INTERVENTIONS:
Device: StatSeal — Patients randomly assigned to the experimental group will have a Statseal Advance (SSA) disc applied after withdrawing the radial sheath 2-4 cm. A Tegaderm dressing will be applied to secure the disc position. The TR band will be applied over the SSA disc with the center of the balloon (the green dot) over the center of the SSA disc. The TR band will be inflated with 8cc of air (which is typically occlusive pressure), and the sheath removed. No deflation will occur immediately. After 20 minutes of pressure, 3 cc of air will be removed from the TR band. After an additional 20 minutes (40 minutes after procedure), the TR band will be completely deflated, and the TR band left in place. After an additional 20 minutes (60 minutes after procedure) the TR band will be removed.
  Other Names: potassium ferrate disc with topical hydrophilic polymer
  Arms: Statseal with TR Band
Device: TR Band — Patients randomly assigned to the control group will have a TR band applied over the arteriotomy site and inflated with 15-18ml of air. After aspirating and clearing the contents of the sheath, the radial sheath will be removed. The TR band will be deflated until bleeding occurs, and 2 ml of air will be reintroduced to provide hemostasis. Patent hemostasis will be documented with plethysmography and oximetry as described below within 5 minutes after band application and removal, and within 30 min of discharge or after 24 hours. The TR band will be left inflated and in place for 2 hours following the procedure for all patients (regardless of diagnostic or PCI procedure), after which deflation attempts will commence.
  Other Names: Hemostasis device
  Arms: TR Band Only

SUMMARY:
The primary objectives of this study are to evaluate the performance of StatSeal Advanced used in conjunction with the TR Band (SSA) as compared to the TR Band without SSA (TRB) relative to: the incidence of peri-procedural radial artery occlusion (RAO) at discharge or 24 hours, whichever occurs first, and the Time to Hemostasis (TTH).

DETAILED DESCRIPTION:
This study is a physician initiated, prospective, observational, two arm, randomized study to be performed at up to four experienced 'Radial First' centers (UCSD, UCLA. Arkansas Heart Hospital and LBVA). A maximum of 180 patients having undergone successful radial catheterization will be enrolled in the study, 60 in each arm. 60 patients will be enrolled at the LBVA. Enrollment will continue at each site on discretion of the investigators until each center enrolls a minimum of 30 patients, or a maximum of 180 patients are enrolled. Clinicians will perform the catheterization in accordance with local standard practice, with a minimum of 5,000 units of unfractionated heparin for anticoagulation. At the start of the TRA procedure, prior to radial artery cannulation, a baseline Pleth-ox exam will be performed for all patients and recorded on the CRF. Ulnar compression will be applied to confirm that the radial artery is patent. Patients with a type D pattern exam will be excluded from the study. At the conclusion of a successful transradial procedure, the patient will be randomized to either SSA or TRB, each device applied per protocol & IFU. It is hypothesized that if radial artery compression time can be shortened to 40 minutes or less, the following could result: improved catheterization lab efficiency, greater patient satisfaction and lower complication rates, including RAO, may be improved.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing diagnostic angiography or PCI via the radial artery
* Patients with a Barbeau test prior to the procedure showing pattern A,B,or

Exclusion Criteria:

* Use of a radial sheath larger than 6 Fr (a 7Fr-in-6 Glidesheath Slender ® is allowed).
* Use of an anticoagulant other than unfractionated heparin or bivalirudin.
* Any anticipated need for continued anticoagulation post-catheterization. Glycoprotein inhibitors are acceptable.
* Any active treatment with oral anticoagulants continued during course of procedure.
* Presence of arteriovenous dialysis fistula in the ipsilateral arm.
* Any physical deformity or trauma / injury of either wrist that would prevent proper placement or function of the hemostasis band.
* Raynaud's syndrome or known peripheral vascular disease of the forearm.
* Mental incompetence or inability to follow the instructions to complete the study.
* History or presence of Radial Artery Occlusion.
* Barbeau test showing Pattern D.
* Patients undergoing catheterization from the femoral or ulnar artery approach.
* Cardiogenic shock or any clinical instability as assessed by the physician performing the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold H Seto, M.D., Principal Investigator — VA Long Beach Hospital
Locations (1):
- Veteran Affairs Long Beach, Long Beach, California, United States

REFERENCES:
- [Result] Seto AH, Rollefson W, Patel MP, Suh WM, Tehrani DM, Nguyen JA, Amador DG, Behnamfar O, Garg V, Cohen MG. Radial haemostasis is facilitated with a potassium ferrate haemostatic patch: the Statseal with TR Band assessment trial (STAT). EuroIntervention. 2018 Dec 7;14(11):e1236-e1242. doi: 10.4244/EIJ-D-18-00101. PMID 29769165
- See also: HTML link to document — https://eurointervention.pcronline.com/article/radial-haemostasis-is-facilitated-with-a-potassium-ferrate-haemostatic-patch-the-statseal-with-tr-band-assessment-trial-stat

RESULTS

PARTICIPANT FLOW:
Groups:
- TR Band Only: Patients randomly assigned to the control group will have a TR band applied over the arteriotomy site and inflated with 15-18ml of air. After aspirating and clearing the contents of the sheath, the radial sheath will be removed. The TR band will be deflated until bleeding occurs, and 2 ml of air will be reintroduced to provide hemostasis. Patent hemostasis will be documented with plethysmography and oximetry as described below within 5 minutes after band application and removal, and within 30 min of discharge or after 24 hours. The TR band will be left inflated and in place for 2 hours following the procedure for all patients (regardless of diagnostic or PCI procedure), after which deflation attempts will commence.
- Statseal With TR Band: Patients randomly assigned to the experimental group will have a Statseal Advance (SSA) disc applied after withdrawing the radial sheath 2-4 cm. A Tegaderm dressing will be applied to secure the disc position. The TR band will be applied over the SSA disc with the center of the balloon (the green dot) over the center of the SSA disc. The TR band will be inflated with 8cc of air (which is typically occlusive pressure), and the sheath removed. No deflation will occur immediately. After 20 minutes of pressure, 3 cc of air will be removed from the TR band. After an additional 20 minutes (40 minutes after procedure), the TR band will be completely deflated, and the TR band left in place. After an additional 20 minutes (60 minutes after procedure) the TR band will be removed.
Period: Overall Study
Arm/Group | TR Band Only | Statseal With TR Band
Started | 90 | 94
Completed | 87 | 93
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TR Band Only | Statseal With TR Band | Total
Number analyzed (Participants) | 87 | 93 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 38 | 73
  >=65 years | 52 | 55 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (9.8) | 65.8 (11.8) | 66.15 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 69 | 71 | 140
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 87 | 93 | 180
Barbeau Class A [Count of Participants; unit: Participants] — A Barbeau test is performed to evaluate the patency of the radiopalmar arch. This is performed by compressing the radial artery for up to 2 minutes and observing the resulting waveform changes. The procedure can be performed in patients with Barbeau classification waveform A, B, or C. All patients received baseline assessment of the hand circulation using the Barbeau's test on a scale A-D, A being patent radial artery. Patients who exhibit a type D waveform indicates an incomplete palmar arch.
  Participants | 76 | 79 | 155

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis Using the Hemostasis Management System (HMS)
Description: Time to deflation for removal of the TR Band (or TR Band and Statseal) for each group was measured in minutes.
Time Frame: within 30 min of discharge or after 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TR Band Only | Statseal With TR Band
Number analyzed (Participants) | 87 | 93
minutes | 160 (42.75) | 42.95 (13.91)

2. Secondary Outcome: Percent of Patients With Radial Artery Occlusion(RAO)
Description: Radial artery occlusion was monitored for all participants using Barbeau's test and pulse oximetry.
Time Frame: within 30 min of discharge or after 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | TR Band Only | Statseal With TR Band
Number analyzed (Participants) | 87 | 93
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: All participants in both groups were monitored post-cardiac catheterization until discharge. Discharge time varied per participant. Outpatient discharge time ranged from two to four hours (unless admitted as inpatient post-procedure). Inpatients were monitored until radial artery patency was observed post-procedure, and were observed for one to two days.
Description: All participants were monitored for radial artery occlusion as well as hematoma formation, and were reported if observed.
Arm/Group | TR Band Only | Statseal With TR Band
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/93
Other Adverse Events (participants affected / at risk) | 9/87 | 18/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TR Band Only (N=87) | Statseal With TR Band (N=93)
Radial Artery Occlusion (Blood and lymphatic system disorders) | 0 | 2 — Radial artery occlusion occurred in 2% of patients in the PFHP group, compared to none in the TRB group.
Hematoma (Blood and lymphatic system disorders) | 9 | 16 — Hematomas in two TRB and three PFHP patients occurred proximal to the TRB early during compression, indicating potentially inaccurate placement of the TR band over the arteriotomy or wire perforation of a small branch during initial access.

LIMITATIONS AND CAVEATS:
The study was not adequately powered for RAO/hematomas, and was open-label so could not be blinded. Our primary endpoint of time to TRB deflation was subject to differential treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT03028025/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03028025/SAP_001.pdf